CLINICAL TRIAL: NCT06942000
Title: Efficacy of Dexmedetomidine as Adjuvant to Intrathecal Bupivacaine in Decreasing Incidence of Post-spinal Shivering in Pregnant Women Undergoing Cesarean Section.
Brief Title: Intrathecal DEX With Bupivacaine Inpost-spinal Shivering After CS.
Acronym: DEX
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Mahmoud, Lecturer of anesthesia, intensive care and pain management, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MSC/AZAST/API029/2/239/1/2025.
Record Dates: First submitted 2025-04-08; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Post Spinal Anesthesia Shivering
Keywords: Cesarean Section; Dexmedetomidine; Intrathecal Anesthesia; Shivering
MeSH Terms: interventions — Dexmedetomidine; Population Groups; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: parturients will be randomly assigned into three equal groups (40 parturients for each group). According to the random number generated by computer, parturient were randomly allocated into three equal groups (40 parturients for each group) to receive either dexmedetomidine 3mcg, dexmedetomidine 5mcg or normal saline in combination with bupivacaine. The randomization sequence was placed in serially numbered opaque envelopes. Before the start of spinal anesthesia, an anesthesiologist who would not involve in the study will prepare relevant drugs according to the randomization sequence.
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group D3: (dexmedetomidine 3mcg group) (Active Comparator): parturients will receive spinal anesthesia consisting of 2ml (10mg) of 0.5% hyperbaric bupivacaine .
  Interventions: Drug: dexmedetomidine 3mcg group
- Group D5: (dexmedetomidine 5mcg group) (Active Comparator): parturients will receive spinal anesthesia consisting of 2ml (10mg) of 0.5% hyperbaric bupivacaine .
  Interventions: Drug: dexmedetomidine 5mcg
- Group C: (Control group) (Placebo Comparator): parturients will receive spinal anesthesia consisting of 2 ml (10 mg) of 0.5% hyperbaric bupivacaine.
  Interventions: Drug: preservative-free 0.9% saline.

INTERVENTIONS:
Drug: dexmedetomidine 3mcg group — 3mcg of preservative-free dexmedetomidine in (0.5 ml) preservative-free 0.9% saline.
  Arms: Group D3: (dexmedetomidine 3mcg group)
Drug: dexmedetomidine 5mcg — 5mcg of preservative-free dexmedetomidine in (0.5 ml) preservative-free 0.9% saline.
  Arms: Group D5: (dexmedetomidine 5mcg group)
Drug: preservative-free 0.9% saline. — (0.5 ml) preservative-free 0.9% saline
  Arms: Group C: (Control group)

SUMMARY:
This prospective, randomized, double-blind, placebo-controlled study to determine whether intrathecal dexmedetomidine, administered along with hyperbaric bupivacaine for covering Cesarean delivery decreases the incidence of shivering associated with spinal anesthesia

DETAILED DESCRIPTION:
The study will be carried out at AL Azhar University Hospitals (Assiut) on 120 parturients belonging to ASA physical status I and II undergoing an elective cesarean delivery under spinal anesthesia procedure.

Sample size was determined by department of statistics of faculty of medicine, Al-Azhar university (Assiut).

Randomization, blinding and allocation concealment parturients will be randomly assigned into three equal groups (40 parturients for each group). According to the random number generated by computer, parturient were randomly allocated into three equal groups (40 parturients for each group) to receive either dexmedetomidine 3mcg, dexmedetomidine 5mcg or normal saline in combination with bupivacaine. The randomization sequence was placed in serially numbered opaque envelopes. Before the start of spinal anesthesia, an anesthesiologist who would not involve in the study will prepare relevant drugs according to the randomization sequence

ELIGIBILITY:
Inclusion Criteria:

* Full-term pregnant women undergoing elective cesarean section under spinal anesthesia.
* singleton pregnancy
* Age: 20 ~ 40 years;
* ASA physical status II ~ III;

Exclusion Criteria:

* parturient less than 20 years and more than 40 years.
* History of uncontrolled comorbidities, cardiac (e.g., pre-eclampsia and hypertension), respiratory, renal or hepatic disease.
* parturients who had allergy to any medication in the study.
* parturients with contraindications to spinal anesthesia (coagulation disorder, infection at site of puncture, raised intracranial tension or any spine deformity)
* parturient who has history of alcohol intake.
* parturient received any medication likely to affect thermoregulation or Veno dilation.
* Refusing to sign informed consent.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Full-term pregnant women
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
efficacy on the incidence and severity of shivering associated with spinal anesthesia. | Shivering will be measured at the following time points: (Immediately after spinal anesthesia, and at 5, 10, 15, 20, 30, 40, 50, 60 and 90 minutes later
  evaluate the effect of intrathecal dexmedetomidine, administered as an adjunct to hyperbaric bupivacaine for Cesarean delivery, on the incidence and severity of shivering associated with spinal anesthesia.

SECONDARY OUTCOMES:
incidence of adverse effects | Immediately after spinal anesthesia, and within 90 minutes later
  the incidence of adverse effects, including nausea, vomiting, bradycardia, hypotension and sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Osama H. Ahmed, MD, Study Director — Professor at Faculty of Medicine, Al-Azhar University, Assiut, Egypt
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Al-Azhar University, Assiut, Egypt, Asyut
  - Mohamed Ali Mahmoud, Asyut

IPD SHARING:
Plan to Share IPD: No
Data is available with corresponding author on reasonable request